CLINICAL TRIAL: NCT00310869
Title: Adolescents Born Preterm: Nurtured Beginnings
Brief Title: Adolescents Born Preterm; Nurtured Beginnings
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Active, not recruiting
Sponsor: Boston Children's Hospital (Other)
Responsible Party: Principal Investigator, Heidelise Als, Professor of Psychology, Boston Children's Hospital
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Prevention
Other Study IDs: 05-02-021
Record Dates: First submitted 2006-04-03; First posted 2006-04-05 (Estimated); Last update posted 2017-06-28 (Actual); Status verified 2017-06

CONDITIONS: Preterm Birth
Keywords: Preterm Birth; Prematurity; NIDCAP; Adolescence; Developmental Care; Follow-up; Neurobehavior
MeSH Terms: conditions — Premature Birth

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- E (Experimental)
  Interventions: Behavioral: Individualized Developmental Care in the NICU

INTERVENTIONS:
Behavioral: Individualized Developmental Care in the NICU — Newborn Individualized Developmental Care and Assessment Program (NIDCAP) utilizes close observation of each infant's thresholds of moving from organization to disorganization and stress, as exhibited by the infant's behavior. Care and environment are then continuously and dynamically adjusted to increase the infant's self-regulation and organization and decrease the infant's stress. This individualized model of NICU care provides an opportunity to investigate the modifiability of very early born infants' brain function and structure and the possibility of reducing or altogether eliminating the disruption and disturbance of fetal brain development in the NICU.
  Other Names: NIDCAP

SUMMARY:
This research study is a long-term follow-up to an earlier study of developmental care. For that study, high risk preterm newborns were randomly assigned to a standard care group, which received the standard care offered in the Newborn Intensive Care Unit (NICU) at the time, or to an experimental group, which received regular behavioral observations to determine if changes in their environment or care were needed. The purpose of the current study is to assess the functioning of these infants again, now that they are adolescents and to compare the groups to determine if the developmental care used in the original study is effective long-term.

DETAILED DESCRIPTION:
The study will test continued long-term intervention effectiveness into adolescence of very early born US preterm infants, who participated in a randomized Newborn Individualized Developmental Care and Assessment Program (NIDCAP) trial, conducted by the principal investigator, while the infants were cared for in the NICU for the first three months after their very premature births. All adolescents to be studied participated as newborns and were assigned either to control care (standard NICU care available at the time), or to experimental care (NIDCAP developmental care, with weekly bedside observations and with daily NIDCAP developmental specialist support to parents and staff), from NICU admission until 2 weeks (w) after expected full-term due date ('corrected' age [CA]).

The strongly brain-based theory underlying the approach to earliest intervention described here has been tested in several experimental studies, which are designed to investigate the effects of planned purposeful modification of experience for very early born infants, who spend the third trimester of gestation in the NICU. NIDCAP is based on an approach which utilizes close observation of each infant's thresholds of moving from organization to disorganization and stress, as exhibited by the infant's behavior. Care and environment are then continuously dynamically adjusted, with the goal to increase the infant's self-regulation and organization and decrease the infant's stress. This individualized model of NICU care provides an opportunity to investigate the modifiability of very early born infants' brain function and structure and the possibility of reducing or altogether eliminating the disruption and disturbance of fetal brain development in the NICU. The randomized scientific trials to date, conducted by the PI and by independent investigators at other settings after formal training show consistent significant neurobehavioral and neurophysiological improvements for the experimental groups across sites and studies.

All the adolescents to be studied were evaluated comprehensively at 2wCA and 9 months (m) CA in terms of not only the commonly measured demographic, medical background and severity of illness variables, but more importantly in terms of comprehensive neurobehavioral and EEG outcome measures, analogues of later developmental competence and disability.

The design of the current study of adolescents is that of a randomized controlled trial (RCT) with two parallel groups (control and experimental), with the question of the independent variable 'group effect' on two dependent measures (adolescent physical growth and cognitive development). In addition to group status, the contribution of four additional independent measures on outcome will also be evaluated: Parent socioeconomic status, parent cognitive function, adolescent physical function and adolescent psychosocial function. The outcome examiners will be blind to subject group status throughout. The design assures a true experimental test of the NICU intervention effects in adolescence.

The significance and importance of the study lays in the unique opportunity to evaluate comprehensively in adolescents the long-term neurodevelopment, learning and adaptive outcomes due to developmental care intervention received in the earliest stage of development. This will be the first study to test the long-term effectiveness of modification of experience in the NICU in a brain-protective, learning-enhancing model for very high-risk, very early-born preterm infants. The importance of the study lies in its potential to contribute significantly to the understanding of preterm brain development in relationship to long-term mental and adaptive functional outcomes in adolescence for the highly jeopardized and growing group of very preterm children. The results are expected to be of key importance in decision and policy development for the evidence-based targeting of sparse special education resources.

ELIGIBILITY:
Inclusion Criteria (when recruited as newborns):

* Gestational age at birth ≤ 28 weeks
* Birth weight ≤ 1250 grams
* In need of mechanical ventilation for at least 24 of the first 48 hours
* Singleton
* Born at the study hospital
* Free of known genetic or acquired infections or abnormalities
* Mother living in the vicinity of the study hospital
* Mother comfortable with English
* Mother free of major physical and mental illnesses

Exclusion Criteria (when recruited as newborns):

* Gestational age at birth > 28 weeks
* Birth weight > 1250 grams
* No mechanical ventilation for the first 48 hours
* Multiple (twin, triplet)
* Not born at the study hospital
* Genetic or acquired infections or abnormalities
* Mother lived outside the vicinity of the study hospital
* Mother was not comfortable with English
* Mother had major physical and/or mental illnesses

Ages: 14 Years to 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Enrollment: 70 (Estimated)
Dates: Start 2005-01 (Actual); Primary Completion 2019-06 (Estimated); Study Completion 2019-12 (Estimated)

PRIMARY OUTCOMES:
Adolescent Cognitive Function | At time of study

SECONDARY OUTCOMES:
Parent socioeconomic status | From birth to time of study
Parent cognitive function | At time of study

CONTACTS AND LOCATIONS:
Overall Officials: Heidelise Als, PhD, Principal Investigator — Boston Children's Hospital
Locations (1):
- Children's Hospital Boston, Boston, Massachusetts, United States

REFERENCES:
- [Background] Als H, Lawhon G, Brown E, Gibes R, Duffy FH, McAnulty G, Blickman JG. Individualized behavioral and environmental care for the very low birth weight preterm infant at high risk for bronchopulmonary dysplasia: neonatal intensive care unit and developmental outcome. Pediatrics. 1986 Dec;78(6):1123-32. PMID 3786036
- [Background] Als H, Lawhon G, Duffy FH, McAnulty GB, Gibes-Grossman R, Blickman JG. Individualized developmental care for the very low-birth-weight preterm infant. Medical and neurofunctional effects. JAMA. 1994 Sep 21;272(11):853-8. PMID 8078162
- [Background] Buehler DM, Als H, Duffy FH, McAnulty GB, Liederman J. Effectiveness of individualized developmental care for low-risk preterm infants: behavioral and electrophysiologic evidence. Pediatrics. 1995 Nov;96(5 Pt 1):923-32. PMID 7478837
- [Background] Als H, Gilkerson L, Duffy FH, McAnulty GB, Buehler DM, Vandenberg K, Sweet N, Sell E, Parad RB, Ringer SA, Butler SC, Blickman JG, Jones KJ. A three-center, randomized, controlled trial of individualized developmental care for very low birth weight preterm infants: medical, neurodevelopmental, parenting, and caregiving effects. J Dev Behav Pediatr. 2003 Dec;24(6):399-408. doi: 10.1097/00004703-200312000-00001. PMID 14671473
- [Background] Als H, Duffy FH, McAnulty GB, Rivkin MJ, Vajapeyam S, Mulkern RV, Warfield SK, Huppi PS, Butler SC, Conneman N, Fischer C, Eichenwald EC. Early experience alters brain function and structure. Pediatrics. 2004 Apr;113(4):846-57. doi: 10.1542/peds.113.4.846. PMID 15060237